CLINICAL TRIAL: NCT04719637
Title: Clinical Study of an Ultrasound Renal Denervation System in Patients With Heart Failure
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Otsuka Medical Devices Co., Ltd. Japan (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: RDN-19-001
Record Dates: First submitted 2020-12-16; First posted 2021-01-22 (Actual); Last update posted 2024-11-08 (Actual); Status verified 2024-11

CONDITIONS: Chronic Heart Failure
Keywords: Denervation; Renal denervation; Heart failure; Ultrasound; Cardiovascular Diseases
MeSH Terms: conditions — Heart Failure; Cardiovascular Diseases

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- PRDS-001 (Experimental): Renal denervation
  Interventions: Device: PRDS-001 Renal Denervation Ultrasound System

INTERVENTIONS:
Device: PRDS-001 Renal Denervation Ultrasound System — Renal Denervation Ultrasound System
  Other Names: renal denervation

SUMMARY:
The purpose is to evaluate the renal denervation system (PRDS-001) for controlling sympathetic nerve over-activation in patients with heart failure, and for its safety in such patients.

ELIGIBILITY:
Inclusion Criteria :

* Patients aged 18 years or older and younger than 85 years at the time of informed consent
* NYHA (New York Heart Association) class II-III
* More than 6 weeks have passed since onset of acute heart failure or acute exacerbation of chronic heart failure
* Washout rate of MIBG [3 (meta)-iodobenzylguanidine] scintigraphy-cardiac is more than 35%
* Patients having continued treatment of heart failure with the same dosage and administration for 4 weeks before obtaining informed consent

Exclusion Criteria :

* Patients with type1 diabetes mellitus, or uncontrolled type 2 diabetes mellitus (HbA1c: ≥ 8%)
* Patients whose eGFR (estimated glomerular filtration rate) is less than 40 mL/min/1.73 m^2 (estimation formula by Japanese Society of Nephrology)
* Patients with concomitant or previous autoimmune or inflammatory bowel disease
* Patients with a history of serious lung disease
* Patients with a history of heart transplantation or VAD [ventricle-assist device]
* Patients receiving reserpine, tricyclic antidepressants, and labetalol hydrochloride (can be used for up to 5 half-lives before informed consent is obtained)
* Patients being treated for Parkinson's disease or Lewy body dementia
* Patients with a history of any severe cardiovascular event (myocardial infarction, coronary artery bypass graft surgery, acute heart failure requiring hospitalization) or severe cerebrovascular event (stroke, transient ischemic event, cerebrovascular accident, etc.) within 3 months before obtaining informed consent
* Patients with persistent atrial fibrillation
* Patients using active implantable medical devices
* Patients with coronary or carotid artery diseases who were deemed necessary by the principal investigator / sub investigator to undergo surgery or PCI (Percutaneous Coronary Intervention) within 6 months after obtaining informed consent
* Patients with contraindications, unacceptable anaphylactic reactions, or uncontrollable allergies to contrast media
* Female patients who are pregnant or breastfeeding
* Patients whose office blood pressure (systolic) is 100mmHg or lower at the time of screening test

Ages: 18 Years to 84 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1 (Actual)
Dates: Start 2021-08-24 (Actual); Primary Completion 2022-02-16 (Actual); Study Completion 2024-08-07 (Actual)

PRIMARY OUTCOMES:
MIBG-cardiac(washout rate) | 6 months

SECONDARY OUTCOMES:
MIBG-cardiac(early; heart-to-mediastinum ratio (H/M), late: H/M) | 6 months
Anaerobic Threshold assessed by CPX (Cardiopulmonary Exercise Testing) | 6 months
Lowest minute ventilation (VE)/carbon dioxide output (VCO2) assessed by CPX | 6 months
Peak oxygen uptake (peak VO2) assessed by CPX | 6 months
Peak VO2/heart rate assessed by CPX | 6 months
VE-VCO2 slope assessed by CPX | 6 months
Peak respiratory exchange ratio assessed by CPX | 6 months
Peak load assessed by CPX | 6 months
Ramp duration assessed by CPX | 6 months
Urinary noradrenalin concentration | 6 months
NYHA class | 6 months
MIBG-renal (washout rate) | 6 months
MIBG-renal (early: kidney-to-mediastinum ratio (K/M), late: K/M) | 6 months

CONTACTS AND LOCATIONS:
Locations (1):
- Osaka University Hospital, Osaka, Japan